CLINICAL TRIAL: NCT02375451
Title: Effect of Childhood Radioiodine Therapy on Salivary Function
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Ari Wassner, Director, Thyroid Program, Division of Endocrinology, Boston Children's Hospital
Other Study IDs: IRB-P00012399
Record Dates: First submitted 2014-10-03; First posted 2015-03-02 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Xerostomia; Hyperthyroidism; Thyroid Cancer
MeSH Terms: conditions — Xerostomia; Hyperthyroidism; Thyroid Neoplasms | interventions — Iodine-131

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Radioiodine: Patients with a history of childhood treatment with radioiodine will be assessed for symptoms of salivary function and measurement of saliva production. These data will be compared to a normal control group.
  Interventions: Other: Radioiodine
- Control: Patients who are similar in age to those in the Radioiodine group, but who did not recieve I-131 therapy.

INTERVENTIONS:
Other: Radioiodine — We will determine if prior radioiodine treatment in childhood impacts salivary function or symptoms. Radioiodine treatment will have been determined by the patient's medical condition and care (NOT assigned by this research study).
  Groups: Radioiodine

SUMMARY:
Radioiodine (I-131) therapy for thyroid disease is known to decrease salivary function in adult patients. The impact of pediatric I-131 exposure on salivary function is unknown. The investigators goals are to answer this question by measuring salivary gland function before and after I-131 administration in children who receive radioiodine therapy at our hospital for thyroid disease.

DETAILED DESCRIPTION:
Radioiodine (I-131) therapy for thyroid disease is known to decrease salivary function in adult patients. The impact of pediatric I-131 exposure on salivary function is unknown. The investigators goals are to answer this question by measuring salivary gland function before and after I-131 administration in children who receive radioiodine therapy at our hospital for thyroid disease. We will use a Modified Shirmer Test to measure saliva production and a questionnaire to evaluation symptoms of xerostomia.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been treated with radioiodine therapy
* Patients who have never received radioiodine therapy (negative control group)

Exclusion Criteria:

* Non-English speaking subjects will be excluded due to our lack of translation support resources at this time. Of note, participation in our study cannot benefit participants in any way.

Ages: 3 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients who have receive I-131 therapy in childhood for thyroid disease, compared to a control group of patients who have never receive I-131 therapy
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2014-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Salivary function (MST value) | 0 to 50 years after radioiodine treatment
  sterile paper strip is used to measure saliva production (noninvasive testing)
Responses to Dry Mouth Questionnaire | At time of visit up to 4 months thereafter.
  Patient questionnaire/survey

SECONDARY OUTCOMES:
Caries history (number of caries noted in dental records) | 1 year before radioiodine administration to 4 months after study visit.

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States